CLINICAL TRIAL: NCT00207493
Title: The Participant Agreement for Contact Tracing (PACT) Study: Enhancing Partner Notification Services.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3305; R30/CCR 119162
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Chlamydia Infection; Contact Tracing
Keywords: sexually transmitted disease; structural intervention; behavioral intervention
MeSH Terms: conditions — Chlamydia Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Kit enhancement to referral
Procedure: patient referral versus contract referral

SUMMARY:
Patients diagnosed with chlamydial infections (a sexually transmitted disease) are asked to notify their sex partners and tell them to seek medical evaluation. This project tests an enhancement to the materials provided to patients to help convince their partners to seek evaluation against the standard of care, which is a brief notification instruction. The desired outcomes are greater levels of notification by participants of their partners and lower levels of reinfection among participants.

DETAILED DESCRIPTION:
Patients diagnosed with chlamydial infections (a sexually transmitted disease) are asked to notify their sex partners and tell them to seek medical evaluation: patient referral. Rates of actual referral by patients are unknown, but estimates derived from several evaluations suggest somewhere between 30 - 55% of partners are notified and tested (for chlamydia). Current prevalence and yearly rates of infection suggest this level of partner notification and treatment is insufficient to control the disease.

As a program, this project has disseminated notification activities to community health centers that see chlamydial infections, all under the aegis of the awardee (Boston Medical Center). Diagnosis and partner notification can be recorded remotely , but centrally accessed through a secure database. To enhance patient referral effectiveness, this project tests brief instructions to refer (standard of care) against a "kit" containing a specific notification of exposure to chlamydia, an accurate health message about the nature and prognosis of the infection (treated and untreated), options for seeking free or low-cost evaluation and treatment, and a satisfaction survey. A second, crossed condition is pure patient referral against a contract (72 hours to notify, after which study staff will refer cases to public health professionals for notification).

Principal outcomes measured are levels of notification by participants of their partners and levels of reinfection among participants. We also measure psychosocial mediating effects, as well as potential unintended consequences of patient referral: incident partner violence against prevalent (baseline rates) violence, depressed affect

ELIGIBILITY:
Inclusion Criteria:

* Sexually active AND
* 15 years old or older AND at least one of:
* Individuals with genitourinary symptoms requiring empiric treatment for chlamydia, OR
* People who self-report that they have had sex with someone who has been diagnosed with an STD within the past 30 days OR
* Asymptomatic female patients with cervicitis diagnosed via a routine pelvic examination.

Exclusion Criteria:

* Subsequent lab confirmation of no chlamydial infection OR
* Sex partner of previously enrolled person OR
* Fear of violence from partner during notification.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 494
Dates: Start 2000-10; Primary Completion 2005-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
1. Participant reinfection rates
2. Participant notification rates
3. Proportion of partners seeking evaluation

SECONDARY OUTCOMES:
1. Experience of violence attributable to notification
2. Relationship prognosis
3. Depression levels

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hogben, PhD, Principal Investigator — Centers for Disease Control and Prevention; Guillermo Madico, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States